CLINICAL TRIAL: NCT04217512
Title: Possible Protective Effect of Pantoprazole in Cisplatin Induced Nephrotoxicity in Patients With Head and Neck Cancer
Brief Title: Pantoprazole in Cisplatin Nephrotoxicity
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: eman ghoneim
Record Dates: First submitted 2019-12-29; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms | interventions — Pantoprazole; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard hydration alone (Active Comparator): Cisplatin with standard hydration
  Interventions: Other: Standard hydration; Drug: Cisplatin
- Pantoprazole high dose (Active Comparator): Cisplatin with standard hydration with pantoprazole 1.6 mg/kg
  Interventions: Drug: Pantoprazole high dose; Other: Standard hydration; Drug: Cisplatin
- Pantoprazole Low dose (Active Comparator): Cisplatin with standard hydration with pantoprazole 0.6 mg/kg
  Interventions: Drug: Pantoprazole low dose; Other: Standard hydration; Drug: Cisplatin

INTERVENTIONS:
Drug: Pantoprazole low dose — Pantoprazole 0.6 mg/kg
  Other Names: zurcal
  Arms: Pantoprazole Low dose
Drug: Pantoprazole high dose — Pantoprazole 1.6 mg\kg
  Other Names: zurcal, Controloc
  Arms: Pantoprazole high dose
Other: Standard hydration — Standard hydration alone
  Other Names: Hydration
Drug: Cisplatin — Cisplatin

SUMMARY:
Pantoprazole in Cisplatin Nephrotoxicity

DETAILED DESCRIPTION:
Pantoprazole in Cisplatin NephrotoxicityPantoprazole in Cisplatin Nephrotoxicity. Is it protective?

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck cancer

Exclusion Criteria:

* GFR less than 59.
* DM
* Elevated liver enzymes more than 3 fold.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with no renal toxicity | 6 months
  The number of patients with no renal toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Eman M Ghonaim, Msc, Principal Investigator — Demonstrator of Clinical Pharmacy; Sahar El-Haggar, Prof, Principal Investigator — Tanta University; Suzy Goher, Lecturer, Principal Investigator — Tanta University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No